CLINICAL TRIAL: NCT00408499
Title: Phase I/II Study of Erlotinib (TARCEVA) and Cetuximab (ERBITUX) in Advanced Solid Tumors, With Emphasis on Non Small Cell Lung Cancer (NSCLC)
Brief Title: Erlotinib and Cetuximab in Treating Patients With Advanced Solid Tumors With Emphasis on Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000517090; P30CA093373 (NIH); UCDCC-177 (Other: University of California Davis); BMS-4608 (Other: Bristol Myers Squibb); BMS-CA225-261 (Other: Bristol Myers Squibb)
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-01

CONDITIONS: Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib + Cetuximab (Experimental): Daily erlotinib combined with weekly cetuximab
  Interventions: Drug: cetuximab; Drug: erlotinib

INTERVENTIONS:
Drug: cetuximab — Cetuximab will be administered intravenously weekly at the maximum tolerated dose (determined in Phase I portion of the study) on a 28 day cycle. Participants will be in this study for at least 2 cycles (8 weeks). If the evaluations show that this treatment has been effective against the participant's cancer, he/she will continue the therapy.
  Other Names: Erbitux
Drug: erlotinib — Erlotinib will be taken by mouth daily on a 28 day cycle. It is in tablet form. The dose will be determined in Phase I portion of the study. Participants will be in this study for at least 2 cycles (8 weeks). If the evaluations show that this treatment has been effective against the participant's cancer, he/she will continue the therapy.
  Other Names: Tarceva

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving erlotinib together with cetuximab may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of erlotinib and cetuximab and to see how well they work in treating patients with advanced solid tumors or progressive or recurrent stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of erlotinib hydrochloride and cetuximab in patients with advanced solid tumors. (Phase I)
* Determine the efficacy of this regimen, in terms of objective tumor response rate, in patients with advanced non-small cell lung cancer (NSCLC) pre-treated with platinum. (Phase II)

Secondary

* Determine the maximum tolerated dose of this regimen in these patients. (Phase I)
* Determine the efficacy of this regimen, in terms of response rate, in these patients. (Phase I)
* Determine the progression-free and overall survival of patients treated with this regimen. (Phase II)
* Determine the frequency and severity of toxicities of this regimen in these patients. (Phase II)
* Determine epidermal growth factor receptor (EGFR) and K-RAS mutation status. (Phase II)
* Evaluate EGFR protein expression and protein expression of downstream markers (e.g., pMAPK, pAKT, p27, and Ki-67). (Phase II)
* Evaluate the levels of marker proteins (e.g., pMAPK, pAKT, p27, and Ki-67) in buccal cells. (Phase II)
* Determine gene copy number by EGFR fluorescent in situ hybridization (FISH). (Phase II)
* Identify EGFR polymorphisms by analysis of genomic DNA from peripheral blood mononuclear cells. (Phase II)
* Determine if the continued presence or absence of mutant K-RAS tumor DNA correlates with response and/or outcome. (Phase II)

OUTLINE: This is a phase I, dose-escalation study followed by an open-label, phase II study.

* Phase I: Patients receive oral erlotinib hydrochloride once daily on days 1-28 and cetuximab IV over 1-2 hours on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride and cetuximab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which ≥ 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

* Phase II: Patients receive erlotinib hydrochloride and cetuximab at the MTD determined in phase I.

Blood and buccal samples are acquired from patients at baseline and prior to courses 2 and 3. Samples are examined by fluorescent in situ hybridization (FISH), immunohistochemistry, polymorphism analysis, and protein expression assays to assess molecular markers (epidermal growth factor receptor, K-RAS, pMAPK, pAKT, p27 and Ki-67) for biologic effects and predictive response.

After completion of phase I treatment, patients are followed for 30 days or until all toxicities resolve. After completion of phase II treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 62 patients will be accrued for this study

ELIGIBILITY:
Inclusion criteria

* For the phase I portion of the study (completed 10/05/08), patients must have cytologically or histologically proven advanced solid tumors for which there is no standard effective therapy available.
* Any number of prior chemotherapy regimens are allowed for the both the Phase I and Phase II portions
* For the phase II portion patients must have cytologically or histologically proven selected stage IIIB (pleural effusion) or IV NSCLC. Patients with NSCLC that have progressed or recurred after first-line therapy for stage IIIA or IIIB may also be considered.
* Patients must have measurable disease by RECIST criteria for the Phase II portion. Disease in previously irradiated sites is considered measurable if there is clear disease progression following radiation therapy. Patients with evaluable disease (bone metastases, pleural fluid, ascites, etc.) may be included in the phase I portion of the trial (completed 10/08/08).
* Must be 18 years of age or older.
* Patients must have a performance status of 0 -2.
* Patients must have an estimated survival of at least 3 months.
* Any prior chemotherapy must have been completed at least 4 weeks prior to start of treatment. For prior mitomycin chemotherapy a 6-week interval is required. Prior radiation must have been completed at least 2 weeks prior to start of therapy. Patients must have recovered from acute reversible medically significant side effects of prior chemotherapy regimens or radiotherapy to NCI-CTC < grade 1 (excluding alopecia). Prior herceptin is allowed.
* Patients must have adequate renal function as documented by a serum creatinine < 1.5 mg/dl or a calculated creatinine clearance of > 45 ml/min (see protocol Appendix D for formula for calculating creatinine clearance).
* Patients must have adequate liver function as documented by serum bilirubin < 1.5 x ULN. AST must be < 2.5 x institutional upper limit of normal.
* Patients must have a pretreatment granulocyte count of >1500/mm3 and platelet count of >100 000/mm3.
* Patients with asymptomatic treated brain metastasis (surgical resection or radiotherapy) may be included if they are neurologically stable and have been off steroids and anticonvulsants for at least 2 weeks.
* All patients must give voluntary written informed consent.
* Patients must be able to take and retain oral medication.
* Documentation of a negative serum pregnancy test.
* Patients on coumadin should have their INR monitored at least once per week or more frequently depending on the investigator's judgment. There have been some case reports of increased INR when coumadin is co-administered with erlotinib.

Exclusion criteria

* Patients who have received erlotinib, cetuximab, or any other EGFR-directed therapy (excluding herceptin).
* Patients with symptomatic brain metastasis or still requiring steroids and anti-convulsants may not be included.
* For the phase II portion of the study, no other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, and any other cancer from which the patient has been disease-free for over five years
* Patients with acute hepatitis or known HIV.
* Patients with active or uncontrolled infection.
* Patients with significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Patients with prior severe infusion reaction to a monoclonal antibody.
* Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).
* Pregnant or breastfeeding females as the effects of these drugs on the unborn fetus are unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-08; Primary Completion 2009-04 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Gandara, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 100 mg Erlotinib, 150 mg/m2 Cetuximab
- Dose Level 2: 100 mg Erlotinib, 200 mg/m2 Cetuximab
- Dose Level 3: 100 mg Erlotinib, 250 mg/m2 Cetuximab
- Dose Level 4: 150 mg Erlotinib, 250 mg/m2 Cetuximab
- Phase II- Dose Expansion: Phase II dose expansion at determined MTD
Period: Phase 1: Dose Levels 1-4
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II- Dose Expansion
Started | 4 | 7 | 3 | 6 | 0
Completed | 2 | 5 | 2 | 6 | 0
Not Completed | 2 | 2 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0
Period: Phase II- MTD Expansion
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II- Dose Expansion
Started | 0 | 0 | 0 | 0 | 44
Completed | 0 | 0 | 0 | 0 | 24
Not Completed | 0 | 0 | 0 | 0 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 9
Not completed — Death | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5
Not completed — treatment delay | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib + Cetuximab
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 32
Age, Continuous [Mean (Full Range); unit: Years] | 62.91 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 54
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing a DLT
Description: Patients will be followed during cycle 1 for the occurrence of a protocol defined dose limiting toxicity
Time Frame: baseline through cycle 1 of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 4 | 7 | 3 | 6
Participants | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Dose Level 1 vs Dose Level 2 vs Dose Level 3 vs Dose Level 4; Test type: Other — Maximum tolerated dose was derived from toxicity data obtained from dose level 1-4; Maximum tolerated dose = 4 — Maximum tolerated dose was determined to be dose level 4: 150 mg Erlotinib, 250 mg/m2 Cetuximab

2. Primary Outcome: Number of Patients Correlated With Best Overall Response.
Description: To determine the efficacy, as measured by objective tumor response rate (RICIST criteria), of daily oral erlotinib and weekly intravenous cetuximab in patients with advanced NSCLC. Best overall response per patient will be reported below.
Time Frame: Every two cycles from first dose to last dose of study drugs
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib + Cetuximab
Number analyzed (Participants) | 64
Participants
  Complete/Partial response | 2
  Stable Disease | 19
  Progressive disease | 22
  Not evaluable | 21

3. Secondary Outcome: Patient Outcome
Description: In the Phase II portion of the study, patients will be followed for both disease free progression by capturing disease progression date and for over all survival by capturing death date.
Time Frame: Patients will be followed until death
Population: 44 patients were enrolled into the Phase II portion of the study
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Expansion: 44 Patients at dose level 4 phase II expansion: 150 mg Erlotinib, 250 mg/m2 Cetuximab
Arm/Group | Phase II Expansion
Number analyzed (Participants) | 44
Participants
  Deceased | 29
  Not followed | 9
  Withdrew consent | 4
  Alive when study terminated | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected day 1 of every cycle for enrolled patients. Total time of collection for all patients: 6 years.
Arm/Group | Erlotinib + Cetuximab
Serious Adverse Events (participants affected / at risk) | 4/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Cetuximab (N=64)
Vomiting (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Thrombosis/thrombus/embolism (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 1
Bronchospasm (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Cetuximab (N=64)
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase Increased (Investigations) | 18
Anorexia (Gastrointestinal disorders) | 7
Bilirubin increased (Investigations) | 13
Acneiform rash (Skin and subcutaneous tissue disorders) | 43
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine Increased (Investigations) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Diarrhea (Gastrointestinal disorders) | 25
Dizziness (Nervous system disorders) | 5
Alkaline phosphatase increased (Investigations) | 9
Dry Skin (Skin and subcutaneous tissue disorders) | 21
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 31
Fever (General disorders) | 4
Headache (Nervous system disorders) | 6
Heartburn (Gastrointestinal disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 13
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 27
Hyponatremia (Metabolism and nutrition disorders) | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 21
Mucositis (Gastrointestinal disorders) | 12
Nail Changes (Skin and subcutaneous tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash NOS (Skin and subcutaneous tissue disorders) | 19
Rash desquamtion (Skin and subcutaneous tissue disorders) | 10
Vomiting (Gastrointestinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes